CLINICAL TRIAL: NCT04789785
Title: : Determining Gastric Emptying Time In Elderly Using Ultrasound Associated With Preoperative Fasting Time
Brief Title: Gastric Emptying Time After Turkish Breakfast
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, SİBEL BEKTAŞ, director, Gaziosmanpasa Research and Education Hospital
Other Study IDs: 182
Record Dates: First submitted 2021-02-22; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Fasting
Keywords: gastric content; gastric ultrasonography; preoperative fasting
MeSH Terms: conditions — Fasting | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound — observation with usg

SUMMARY:
DETERMINING GASTRIC EMPTYING TIME IN ELDERLY USING ULTRASOUND ASSOCIATED WITH PREOPERATIVE FASTING TIME

Background:

Gastric contents aspiration is the most crucial complication of general anaesthesia. There are limited studies to assess the gastric volume ultrasound to clarify an appropriate fasting time before surgery. Gastric content will examine after a traditional Turkish breakfast with ultrasound.

Methods:

After the first ultrasound examination by asking 8 hours fasting ,gastric emptying time(GET) was determined by serial gastric ultrasound examinations with two ultrasonographers and GET identified by real time USG evaluations in every 1 hour.

All ultrasound assessments on volunteers will made both in the supine position and right lateral decubitus (RLD) from the epigastric area by using a convex probe.

This study is the first one which examine gastric emptying time after a standard Turkish breakfast in over 65 years Turkish population by measuring antral cross section area (CSA) using noninvasive ultrasound.

DETAILED DESCRIPTION:
Preoperative fasting has always been problematic in preoperative patients because of the pulmonary aspiration hazard and discomfort of prolonged fasting. Although stomach scintigraphy has been accepted as a gold standard for imaging method of evaluating gastric content; recently, ultrasound is being a simple, efficient, available and non invasive alternative. Preoperative fasting is especially difficult in elderly because of comorbidities, dehydration, drug therapies. Therefore, in this study gastric emptying time will be identified after a standard Turkish breakfast in over 65 years old Turkish population to clarify fasting time, measuring antral cross section area (CSA) by using non invasive ultrasound for the first time. Ultrasound assessments on volunteers will be made both in the supine position and right lateral decubitus (RLD) from the epigastric area by using a convex probe. After visualization of gastric antrum according to landmarks such as abdominal aorta, superior mesenteric artery and the left lobe of liver; antrum will measured in two sagittal planes: craniocaudal (CC) and anteroposterior(AP) diameters. Gastric emptying time will be identify by real time usg done by 1 hour intervals.This is the first study with ultrasound evaluation of gastric emptying time in Turkish population after a traditional Turkish breakfast.

ELIGIBILITY:
Inclusion Criteria:

* over 65 years of age who have not any comorbidities

Exclusion Criteria:

* gastrointestinal and functional disorders, previous oesophageal or upper abdomen surgery.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: over 65 years of age Turkish volunteers without comorbity
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
evaluating gastric emptying time assosiated with preoperative fasting | base and real time measurements for 6 hours by 1 hour intervals
  By measuring gastric cross section area using ultrasound to find the emptying time about 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa TREH, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Publishing in a journal

REFERENCES:
- [Background] Soenen S, Rayner CK, Horowitz M, Jones KL. Gastric Emptying in the Elderly. Clin Geriatr Med. 2015 Aug;31(3):339-53. doi: 10.1016/j.cger.2015.04.003. Epub 2015 May 11. PMID 26195094
- [Background] Bolondi L, Bortolotti M, Santi V, Calletti T, Gaiani S, Labo G. Measurement of gastric emptying time by real-time ultrasonography. Gastroenterology. 1985 Oct;89(4):752-9. doi: 10.1016/0016-5085(85)90569-4. PMID 3896910